CLINICAL TRIAL: NCT01931761
Title: A Phase I, Single-centre, Non-randomised, Open-label, Pharmacokinetic and Mass Balance Study of Orally Administered [14C]-Selumetinib in Healthy Male Volunteers
Brief Title: Study Evaluating Absorption, Distribution, Metabolism and Excretion (ADME) of Single Dose [14C] Selumetinib in Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: D1532C00077
Record Dates: First submitted 2013-08-27; First posted 2013-08-29 (Estimated); Last update posted 2015-06-30 (Estimated); Status verified 2015-06

CONDITIONS: Solid Tumours
Keywords: Pharmacokinetics, mass balance, AZD6244
MeSH Terms: interventions — Carbon-14; AZD 6244

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- [C14] selumetinib 75mg single dose (Experimental): [C14] selumetinib 75mg single dose
  Interventions: Drug: [C14] selumetinib (oral)

INTERVENTIONS:
Drug: [C14] selumetinib (oral) — Single oral administration [C14] 75mg
  Other Names: Selumetinib

SUMMARY:
To evaluate the absorption, distribution, metabolism and excretion (ADME) of single dose [14C] selumetinib in volunteers

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated, written informed consent prior to any study specific procedures.
* Have a body mass index (BMI) between 18 and 32 kg/m2 inclusive and weigh at least 50 kg and no more than 100 kg, inclusive.
* Regular bowel movements (ie, on average production of at least 1 stool per day).

Exclusion Criteria:

* Current or past history of central serous retinopathy or retinal vein thrombosis, intraocular pressure greater than 21 mmHg or uncontrolled glaucoma.
* Exposure to radiation levels above background exceeding 5 mSv in the last 12 months or 10 mSv in the last 5 years.
* History or presence of any clinically significant disease or disorder in the opinion of the investigator
* Any clinically important abnormalities in clinical chemistry, haematology, or urinalysis results, vital signs or ECG at baseline in the opinion of the Investigator.

Ages: 50 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2013-10; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Concentration of total radioactivity in blood and plasma and percentage of radioactive dose in urine and faeces and total balance | Samples collected prior to treatment, during treatment and follow-up for a maximum of 14 days

SECONDARY OUTCOMES:
Metabolite profiling and identification in plasma and excreta | Samples collected prior to treatment, during treatment and follow-up for a maximum of 14 days.
Pharmacokinetic parameters of selumetinib | Samples collected prior to treatment, during treatment and follow-up for a maximum of 14 days.
  Cmax, tmax, t½, AUC, CL/F, Vz/F, MRT, fe, Ae, CLR
Plasma concentrations of selumetinib | Samples collected prior to treatment, during treatment and follow-up for a maximum of 14 days
Safety | Assessments prior to treatment and after treatment including follow up.
  Adverse events, vital signs, electrocardiogram, haematology, clinical chemistry, urinalysis, physical examination, left ventricular ejection fraction, and opthalmology assessments.

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Mair, MD, Principal Investigator — University of Aberdeen
Locations (1):
- Research Site, Ruddington, United Kingdom

REFERENCES:
- [Derived] Dymond AW, Howes C, Pattison C, So K, Mariani G, Savage M, Mair S, Ford G, Martin P. Metabolism, Excretion, and Pharmacokinetics of Selumetinib, an MEK1/2 inhibitor, in Healthy Adult Male Subjects. Clin Ther. 2016 Nov;38(11):2447-2458. doi: 10.1016/j.clinthera.2016.09.002. Epub 2016 Oct 15. PMID 27751676
- See also: CSR_Synopsis_D1532C00077.pdf — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1869&filename=CSR_Synopsis_D1532C00077.pdf